CLINICAL TRIAL: NCT06947408
Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of IBI3002 Multiple Dosing in Healthy Participants and Patients With Asthma - A Randomized, Double-Blind, Placebo-Controlled, Dose-Ascending Study
Brief Title: A Study to Evaluate the Safety and Tolerability of Multiple Dose of IBI3002 in Healthy and Asthmatic Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI3002A102
Record Dates: First submitted 2025-04-10; First posted 2025-04-27 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part B IBI3002 900mg SC (Experimental): Patients with asthma will receive IBI3002 900mg SC at Week 0, 2, 4, 6, 8 and 10
  Interventions: Drug: IBI3002
- Part B Placebo (Placebo Comparator): Patients with asthma will receive matched placebo
  Interventions: Drug: Placebo
- Part A IBI3002 300mg SC (Experimental): Healthy Participants will receive IBI3002 300mg SC at Week 0, 2, 4, and 6
  Interventions: Drug: IBI3002
- Part A IBI3002 600mg SC (Experimental): Healthy Participants will receive IBI3002 600mg SC at Week 0, 2, 4, and 6
  Interventions: Drug: IBI3002
- Part B IBI3002 300mg SC (Experimental): Patients with asthma will receive IBI3002 300mg SC at Week 0, 2, 4, 6, 8 and 10
  Interventions: Drug: IBI3002
- Part A Placebo (Placebo Comparator): Healthy Participants will receive matched placebo
  Interventions: Drug: Placebo
- Part A IBI3002 600mg IV (Experimental): Healthy Participants will receive IBI3002 600mg IV at Week 0, 2, 4, and 6
  Interventions: Drug: IBI3002
- Part A IBI3002 900mg SC (Experimental): Healthy Participants will receive IBI3002 900mg SC at Week 0, 2, 4, and 6
  Interventions: Drug: IBI3002
- Part A IBI3002 150 mg SC (Experimental): Healthy Participants will receive IBI3002 150mg SC at Week 0, 4 and 8
  Interventions: Drug: IBI3002

INTERVENTIONS:
Drug: Placebo — Healthy participants and patients with asthma will receive matched placebo.
  Arms: Part A Placebo; Part B Placebo
Drug: IBI3002 — Healthy participants and patients with asthma will receive IBI3002 at the corresponding dose and dosing interval.
  Arms: Part A IBI3002 150 mg SC; Part A IBI3002 300mg SC; Part A IBI3002 600mg IV; Part A IBI3002 600mg SC; Part A IBI3002 900mg SC; Part B IBI3002 300mg SC; Part B IBI3002 900mg SC

SUMMARY:
This study is a randomized, double-blind, placebo-controlled multiple dose ascending study in healthy participants and patients with asthma. Healthy participants will be enrolled in Part A and patients with asthma in Part B:

1. Part A: 40 healthy participants will be enrolled across 5 cohorts, including dose levels of 150mg, 300mg, 600mg, 900mg SC, and 600mg IV. In each cohort, there will be 8 participants randomized at a ratio of 6:2 to receive IBI3002 or matched placebo. The study consists of a screening period, a double-blind treatment period and a safety follow-up period. The study has a total duration of approximately 12 to 14 weeks.
2. Part B: 20 patients with asthma will be enrolled across 2 cohorts, including dose levels of 300mg and 900mg SC. In each cohort, there will be 10 participants randomized at a ratio of 8:2 to receive IBI3002 or matched placebo. The study consists of a screening period, a double-blind treatment period and a safety follow-up period. The study has a total duration of approximately 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. (Part A and B) The body weight of men ≥ 50kg, and of women ≥ 45kg; Body mass index (BMI) between 18 and 32 kg/m2 (including cut-off values).
2. (Part B) Diagnosed with asthma for at least 12 months according to the Global Initiative for Asthma (GINA) and confirmed by the Investigator.
3. (Part B) Evidence of airway reversibility within 5 years prior to screening, including but not limited to a positive bronchodilation test or bronchoprovocation test. If the historical results are not available, tests during the screening period will also be accepted.
4. (Part B) Medium-high dose ICS therapy (defined as a daily dose of ≥250μg fluticasone propionate or equivalent ICS dose) in combination with at least one second controller [e.g., LABA, LAMA, or LTRA for at least 3 months with a stable dose for at least 1 month prior to randomization.
5. (Part B) Pre-BD FEV1 ≤ 80% of prediction.

Exclusion Criteria:

1. (Part A and B) Diseases that have an impact on the participant's own safety or participation in the study as judged by the investigator. This includes, but not limited to, mental disorders, diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, or metabolic system.
2. (Part A and B) Participants with known history of active tuberculosis or clinical suspicion of tuberculosis (including but not limited to pulmonary tuberculosis, lymph node tuberculosis, tuberculous pleurisy, etc.); or positive T-SPOT.TB during the screening period, or evidence of suspected tuberculosis on chest imaging, or any other clinical evidence of latent tuberculosis.
3. (Part A and B) A history of malignancy, except for localized basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) of the skin that has been resected or cured.
4. (Part B) History of a life-threatening asthma attack requiring mechanical ventilation, and/or an asthma attack related to hypercapnia, respiratory failure, or hypoxic epilepsy within 5 years prior to screening.
5. (Part B) History of an asthma worsening or exacerbation that resulted in an visit to emergency room or hospitalization, or an increase in asthma controller, or requiring any systemic glucocorticoid therapy within 3 months prior to screening.

The above information is not intended to contain all considerations relevant to a participant's potential participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
To evaluate the Incidence of sudden adverse events of healthy participants and patients with asthma receiving IBI3002 multiple ascending doses. | baseline to Week16
  Incidence of adverse events (AEs) and serious adverse events (SAEs) after IBI3002 multiple doses in healthy participants;

SECONDARY OUTCOMES:
To assess PK parameters of healthy participants and patients with asthma receiving IBI3002 multiple ascending doses. | baseline to Week16
  PK parameters include, the maximum concentration (Cmax), after multiple doses.
To assess PK parameters of healthy participants and patients with asthma receiving IBI3002 multiple ascending doses. | baseline to Week16
  PK parameters include, the time to achieve Cmax (Tmax), after multiple doses.
To assess PK parameters of healthy participants and patients with asthma receiving IBI3002 multiple ascending doses. | baseline to Week16
  PK parameters include, the area under the concentration-time curve (AUC) ,after multiple doses.
To assess PK parameters of healthy participants and patients with asthma receiving IBI3002 multiple ascending doses. | baseline to Week16
  PK parameters include the trough concentration (Cmin) after multiple doses.
To assess the incidence of immunogenicity of healthy participants and patients with asthma receiving IBI3002 multiple ascending doses. | baseline to Week16
  the incidence of immunogenicity of IBI3002.

CONTACTS AND LOCATIONS:
Locations (1):
- China-japan Friendship Hosipital, Beijing, Beijing Municipality, China